CLINICAL TRIAL: NCT00646802
Title: Vaginal Progesterone as a Maintenance Treatment in Women With Previous Preterm Labor. Randomized, Double Blinded, Placebo-controlled Trial
Brief Title: Vaginal PROgesterone as Maintenance Treatment After an epISode of prEterm Labor (PROMISE Study)
Acronym: PROMISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Montse Palacio, MD, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROMISE
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Threatened Premature Labor
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Progesterone 200 mg
  Interventions: Drug: Progesterone
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — 1 vaginal capsule, 200 mg, once daily since gestation age 36 weeks and 6 days
  Arms: A
Drug: Placebo — 1 vaginal capsule, once daily since gestational age of 36 weeks and 6 days
  Arms: B

SUMMARY:
Eligible patients will be informed and asked to enroll in the study at hospital admission. A transvaginal ultrasound examination will be performed to determine cervical length. If an eligible woman accepts to participate, patient will be randomized to one of the study arms assigned in a double blind basis. Patient will receive the medication (vaginal capsule of progesterone or placebo). The patient will administer herself one vaginal capsule in a daily basis since gestational age of 36 weeks and 6 days as the primary endpoint is to demonstrate that the use of a maintenance treatment with vaginal progesterone is able to reduce the incidence of preterm birth before 34.0 and 37.0 gestational weeks. After delivery, perinatal and neonatal data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged between 18 - 45 years
* Gestational age between 24.0 and before 33.6 gestational weeks
* Singleton pregnancy
* Patients admitted because of preterm labor who have been successfully treated of any tocolytic drugs (β-mimetics drugs, nifedipine, atosiban)
* Ultrasound cervical length at discharge < 25 mm
* Signed patient consent form (CI)

Exclusion Criteria:

* Known or suspected infection, premature rupture of membranes or any other pathological gravid maternal or fetal condition coexisting at hospital admission (Pre-eclampsia, RCIU) which may induce iatrogenic labor.
* Present or previous liver disease, present or previous cholestasis gravidarum, abnormal hepatic blood tests.
* With known allergy to progesterone or peanuts (excipient).
* Grade 2 (or upper) renal or liver laboratory abnormalities
* Treated from dependent-hormone malignant cancer (i.e., breast carcinoma...)
* With Diabetes mellitus or insulinized gestational diabetes
* Treated with heparin
* Drug abuse
* Inadequate treatment compliance

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 265 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of deliveries before week 34 of gestation | week 34 of gestation

SECONDARY OUTCOMES:
Median time from randomization to delivery | delivery
Ultrasound cervical length | week +5

CONTACTS AND LOCATIONS:
Overall Officials: Montse Palacio, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (12):
- Spain (12):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Institut Universitari Dexeus, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Sant joan de Déu de Manresa, Manresa, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital de Terrassa. CST, Terrassa, Barcelona
  - Hospital de Basurto, Bilbao, Bilbao
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital U Gregorio Marañon, Madrid, Madrid
  - Hospital Virgen de la Macarena, Seville, Seville
  - Hospital Clinico U. Lozano Blesa, Zaragoza, Zaragoza